CLINICAL TRIAL: NCT03583671
Title: Prevalence of Molar Incisor Hypomineralization Among a Group of Egyptian Children Aged From Eight to Twelve Years Old in Dakahlia Governorate: A Cross Sectional Study
Brief Title: Prevalence of Molar Incisor Hypomineralization Among a Group of Egyptian Children From 8 to 12 Years Old in Dakahlia
Acronym: MIH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana Mohamed Mohamed EL-Abassery, Master dental student in Cairo University, Cairo University
Other Study IDs: CEBD-CU-2018-06-22
Record Dates: First submitted 2018-06-22; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor Hypomineralization , enamel defects.
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the prevalence of MIH among a group of Egyptian children aged from 8-12 years old in Dakahlia governorate schools.

DETAILED DESCRIPTION:
* Clinical examination will be carried out in the school laboratory or an empty class, in day light, teeth will be cleaned gently using gauze and wet with saliva during examination. A disposable diagnostic set (mirror, probe) will be used for each patient where mirrors will be used for proper visualization especially for maxillary teeth. Blunt explorers will be used to aid in tactile sensation if needed, as during the differentiation between rough and smooth enamel edges and/or during the inspection of the caries extent if it exists. No diagnostic radiographs will be taken.
* An examination chart (Appendix 1) will be filled for each child including: date, name, age, address, gender, school, medical health and any previous dental treatment, followed by clinical examination to the four first permanent molars and the eight maxillary and mandibular incisors to detect the presence of MIH and its severity based on European Academy of Pediatric Dentistry (EAPD) criteria . To diagnose Molar Incisor Hypomineralization, at least one affected first permanent molar is required. Extracted first permanent molar will be recorded as affected if another first permanent molar has a defecting MIH
* Each child affected with MIH will be given a letter outlining his dental health status, to inform the parents and indicate the need for treatment.

Examination chart

Date:

Personal information:

Name: Age: Gender:

Address:

School:

Medical history:

Dental history:

Clinical examination:

8 7 6 5 4 3 2 1 1 2 3 4 5 6 7 8

8 7 6 5 4 3 2 1 1 2 3 4 5 6 7 8

Severity according to EAPD:

Code Description Severity 0 No defect

1. White or creamy demarcated opacities/mild Mild
2. Yellow or brown demarcated opacities Mild
3. a Enamel loss Moderate

3b Enamel and dentin loss Severe 3c Atypical large cavities extended to pulp and covering one or more tubercle Severe 4 Atypical restorations Severe 5 Extracted tooth Severe

Comments:

MIH: presence / absence Severity: Mild / Moderate /Severe

(Appendix 1)

ELIGIBILITY:
Inclusion Criteria:

* Acceptance for participation in the study.
* Children aged from 8-12 years old.
* Eruption of at four first permanent molars.
* Both genders.

Exclusion Criteria:

* Uncooperative children.
* Children with orthodontic appliances.
* Children with systemic diseases which may affect teeth development.
* Children suffering from any other type of enamel defect as enamel hypoplasia and amelogenesis imperfecta.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Egyptian children aged from 8-12 years old in Dakahlia governorate schools.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Molar Incisor Hypomineralization | 6 months
  measuring method:clinical examination measuring unit: binary method

SECONDARY OUTCOMES:
Severity of Molar Incisor Hypomineralization | 6 months
  measuring method: clinical examination measuring unit:Modified index (based on European Academy of Pediatric Dentistry criteria 2003, 2009)

CONTACTS AND LOCATIONS:
Overall Officials: Soad Abd EL-Moniem, Ass.prof., Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided